CLINICAL TRIAL: NCT03163628
Title: Performance Assessment of 7 Biomarkers for the Diagnosis of Severe Bacterial Infections in Children Aged From 7 Days to 36 Months.
Brief Title: biomArkers to differeNtiate bacTerial From vIral iNfEctions
Acronym: ANTOINE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 69HCL16_0799
Record Dates: First submitted 2017-05-22; First posted 2017-05-23 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Infection, Bacterial; Infection Viral
Keywords: severe bacterial infection; acute infection; infection viral; biomarker combination; diagnostic; child
MeSH Terms: conditions — Bacterial Infections; Virus Diseases; Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 7 biomarkers combination (Experimental)
  Interventions: Biological: Diagnostic performances of a combination of biomarkers

INTERVENTIONS:
Biological: Diagnostic performances of a combination of biomarkers — 3 ml of blood will be drawn at inclusion at the same time of the venipuncture prescribed for standard care. The dosage of the 7 biomarkers will be performed in a central laboratory. The adjudication committee will classify patients in 6 groups, based on their clinical data. The committee will not be aware of the biological results. The analysis of Train Set data will aim to identify the most effective combination of markers in response to the primary objective of identifying biomarkers for the diagnosis of severe bacterial infections. The best combination selected will then be applied to the Test Set data (approximately the other half of patients), in order to obtain its real and unbiased performance.
  The calculation of positive and negative likelihood ratios will be performed.
  The targeted performances are:
  * A positive likelihood ratio (LR +) of 5.67 minimum, ideally greater than 8.5.
  * A negative likelihood ratio (LR-) of 0.5 maximum, ideally less than 0.3.

SUMMARY:
ANTOINE is a prospective trial which aims to assess diagnostic performance of 7 biomarkers for the diagnosis of severe bacterial infections (SBI) in children aged from 7 days to 36 months.

Fever is a frequent cause of consultation in pediatric emergency departments. Clinical diagnostic tools are rare and discrimination between severe bacterial infection and viral infection is difficult to confidently state. The prevalence of severe bacterial infections (IBS) varies from 10 to 25% according to the studies. Biological markers such as procalcitonin (PCT) and C-reactive protein (CRP) are commonly used in clinical practice. These markers have bacterial specificity but share a wide range of values with viral infections and do not make it possible to exclude or to confirm definitively the diagnosis of IBS. The use of new markers to improve the diagnosis of bacterial and viral infections is increasingly studied in adults. The diagnostic value of these new markers has been demonstrated by associating their dosage with that of CRP for example. This is the case for IP-10, TRAIL or MxA. However, very few pediatric studies have been carried out to date on these new biomarkers. However, in pediatrics, these diagnostic tools based on the combination of biomarkers to discriminate against viral and bacterial infections could be a major help in the suspicions of IBS. 7 biomarkers were selected to be evaluated in this study. This study is designed to determine the best biomarkers combination for the SBI diagnosis on a cohort of 800 patients.

ELIGIBILITY:
Inclusion Criteria:

* Febrile children:

  * Between 7 days and 3 months old : fever >38°C for more than 6 hours (late neonatal fever suspected) for which the physician prescribed venipuncture
  * Between 3 months and 36 months old : fever ≥38,5°C for more than 6 hours and less than 7 days for which the physician prescribed venipuncture for suspected severe bacterial infection
* Patient with national health cover
* Consent form signed by at least one parent

Exclusion Criteria:

* Children treated by antibiotherapy within the past 48h
* Children with congenital or acquired immunodeficiency syndrome or long-term immunosuppression treatment
* Vaccinated children within 48h by an inactivated vaccine or within 10 days for the MMR vaccines
* Children with a chronic disease
* undergoing surgery within 7 days before inclusion

Ages: 7 Days to 36 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 983 (Actual)
Dates: Start 2017-06-06 (Actual); Primary Completion 2019-06-12 (Actual); Study Completion 2019-06-12 (Actual)

PRIMARY OUTCOMES:
Diagnosis of severe bacterial infection (SBI) | at Day 7
  Diagnostic performance of the biomarkers combination will be compared to the diagnostic performances of CRP alone and PCT alone, based on the adjudication committee classification (gold standard).
  The Adjudication Committee will sort patients in 6 different groups according to their clinical data: (1) proved SBI, (2) presumed SBI, (3) both viral & bacterial infection, (4) proved viral infection, (5) presumed viral infection, & (6) not classifiable patient. To answer the primary outcome, the SBI class will group proved SBI (1), presumed SBI (2) and both viral & bacterial infection (3).

SECONDARY OUTCOMES:
Diagnosis of viral infection | at Day 7
  Diagnostic performance of the biomarkers combination will be compared to the diagnostic performances of CRP alone and PCT alone, based on the adjudication committee classification (gold standard).
  The Adjudication Committee will sort patients in 6 different groups according to their clinical data: (1) proved SBI, (2) presumed SBI, (3) both viral & bacterial infection, (4) proved viral infection, (5) presumed viral infection, & (6) not classifiable patient. To answer this secondary outcome, the SBI class will group (4) proved viral infection, (5) presumed viral infection.
Unfavorable evolution | at Day 7
  Evaluate the possible association between biomarkers concentration and patient unfavorable evolution, defined as:
  * For hospitalized patient : entry in a health department with an higher level of care or death within 7 days after study inclusion
  * For non-hospitalized patient : hospitalization or death within 7 days after study inclusion

CONTACTS AND LOCATIONS:
Overall Officials: Yves GILLET, MD, Principal Investigator — Hospices Civils de Lyon
Locations (3):
- France (3):
  - Hospices Civils de Lyon, Bron
  - Hôpital Louis Mourier - APHP, Colombes
  - Hôpital Nord Ouest, Gleizé

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Trouillet-Assant S, Viel S, Ouziel A, Boisselier L, Rebaud P, Basmaci R, Droz N, Belot A, Pons S, Brengel-Pesce K, Gillet Y, Javouhey E; Antoine Study Group. Type I Interferon in Children with Viral or Bacterial Infections. Clin Chem. 2020 Jun 1;66(6):802-808. doi: 10.1093/clinchem/hvaa089. PMID 32359149